CLINICAL TRIAL: NCT07248202
Title: A Comparison Between the Effect of Ketamine-lidocaine Versus Ketamine-fentanyl for Induction of Anesthesia on Cerebral Perfusion Guided by Near Infra-red Spectroscopy in Patients With Coronary Artery Disease and Left Ventricular Systolic Dysfunction Undergoing Elective Coronary Artery Bypass Graft Surgery: (A Randomized Controlled Study)
Brief Title: Ketamine-lidocaine Versus Ketamine-fentanyl for Induction of Anesthesia in Patients With Left Ventricular Systolic Dysfunction Undergoing Elective Coronary Artery Bypass
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-396-2024
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease (CAD); Left Ventricular (LV) Systolic Dysfunction; Induction Anesthesia; Coronary Bypass Graft Surgery; Ketamine; Fentanyl; Lidocaine
MeSH Terms: conditions — Coronary Artery Disease | interventions — Fentanyl; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fentanyl group (Active Comparator): fentanyl bolus during induction of anesthesia
  Interventions: Drug: Fentanyl (IV)
- lidocaine group (Active Comparator): lidocaine bolus during the induction of anesthesia
  Interventions: Drug: lidocaine

INTERVENTIONS:
Drug: Fentanyl (IV) — patients will receive 1 mcg/kg of Fentanyl (10 mcg/mL).
  Arms: fentanyl group
Drug: lidocaine — patients will receive 1 mg/kg lidocaine (10mg/mL)
  Arms: lidocaine group

SUMMARY:
There is no consensus on the ideal induction technique for patients with coronary artery disease and left heart dysfunction. Induction for cardiac surgery focuses on maintaining hemodynamic stability, optimizing myocardial oxygen balance, and minimizing the intubation stress response. Ketamine provides stable hemodynamics in patients with impaired ventricular function, though combining it with opioids to blunt the intubation response may increase post-induction hypotension.

Systemic lidocaine has anesthetic-sparing properties and has been shown to potentiate agents such as thiopentone, propofol, and midazolam. The ketamine-lidocaine combination has also demonstrated favorable hemodynamic effects in septic shock.

This study compares ketamine/fentanyl versus ketamine/lidocaine in term of their impact on cerebral perfusion during CABG. No prior data address these effects, and the goal is to identify the induction regimen that better preserves cerebral oxygenation.

DETAILED DESCRIPTION:
Upon arrival to the operating room, initial monitoring will include five lead electrocardiograms, non-invasive blood pressure, and pulse oximetry. At the attending anesthetist's discretion, intravenous midazolam will be administered for anxiolytics. Under local anesthesia, an arterial line will be placed in the radial artery of the non-dominant hand and central venous line will be placed in the right internal jugular vein.

Cerebral oximetry monitoring using Near-Infrared Spectroscopy (NIRS) bilaterally (CASMED, Module series Fore-sight Elite, [SN]1931030) will be applied to all patients. After cleansing of the adjacent skin area with alcohol, an adhesive optode pad was placed over each fronto-temporal area. Resting baseline rSO2 values will be obtained after waiting at least 1 min after placement of sensors once values had stabilized. Bispectral index (BIS) will be applied.

The baseline data for the heart rate, systolic, diastolic, and mean systemic arterial pressures will be recorded from the average ward measurement the day before surgery.

in all patients, ketamine will be injected slowly at 1.5 mg/kg in 0.25 mg/kg increments until clinical loss of consciousness. Clinical loss of consciousness (defined as no response to auditory command) will be assessed by asking the patients repeatedly to open their eyes. After loss of consciousness, atracurium 0.5 mg/kg will be administered to facilitate tracheal intubation. Tachycardia and hypertension, (20% increase heart rate, blood pressure from baseline reading) will be managed by a 50 mcg-bolus of Fentanyl. Anesthesia will be maintained by isoflurane (adjusted to maintain end-tidal minimal alveolar concentration of 1-1.2 %) in oxygen/air mixture. Mechanical ventilation will be adjusted to maintain end-tidal CO2 of 35-40 mmHg Any episode of hypotension (defined as mean arterial pressure [MAP] < 70% of the baseline reading and/or MAP <65mmHg, will be managed by 5 mcg norepinephrine (which could be repeated if hypotension persists for 1-min, NE infusion will be started if persisted after 3 boluses). Ephedrine bolus will be give if hypotension was associated with bradycardia.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease
* with moderate to severe left ventricular dysfunction (ejection fraction < 40%),
* scheduled for elective CABG surgery

Exclusion Criteria:

* associated chronic stroke, TIA , carotid occlusive disease( due to abnormal vasomotor activity), patients with known neurological impairment (cerebral infarction , dementia ), significant carotid artery stenosis ,
* valvular heart disease,
* persistent arrhythmias,
* congestive cardiac failure,
* on mechanical ventilation,
* intra-aortic balloon pump,
* emergency surgery,
* and those with known allergy to any of the study's drugs,
* severe systemic non-cardiac disease and
* patients with baseline NIRS reading < 60%
* Patients with dementia or visual or auditory impairment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
average postinduction NIRS | every 5 min after induction of anesthesia until 20 min after
  average values of NIRS reading after induction of anesthesia

SECONDARY OUTCOMES:
mean arterial pressure | every minute after induction of anesthesia until 20 min after induction
  invasive mean arterial pressure
heart rate | every minute after induction of anesthesia until 20 min after induction
  bpm
NRIS | during induction, 1 min after induction, during intubation, then every 5 minutes for 20 min
  average of left and right side reading
cerebral hypoperfusion | during induction, 1 min after induction, during intubation, then every 5 minutes for 20 min
  NIRS<60% or <90% of baseline reading
hypotension | immediately after induction of anesthesia until 20 min after induction
  mean arterial pressure <70% of baseline or <65 mmHg
extra fentanyl bolus | immediately after induction of anesthesia until 20 min after induction
  mcg
postoperative myocardial infarction | after extubation until 30 days postoperative
  elevated troponin and new ECG changes
postoperative stroke | after extubation until 30 days postoperative
  new neurologic deficit
postoperative acute kidney injury | after extubation until 30 days postoperative
wound infection | after extubation until 30 days postoperative
renal replacement therapy | after extubation until 30 days postoperative

OTHER OUTCOMES:
vasopressor dose | immediately after induction until 20 min after induction

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data related to this research are available form the PI upon reasonable request